CLINICAL TRIAL: NCT01129882
Title: An Open-Label, Multicenter, Rollover, Long-term Study of Aripiprazole Intramuscular Depot in Patients With Schizophrenia
Brief Title: An Open-Label, Multicenter, Rollover, Long-term Study of Aripiprazole Intramuscular Depot in Participants With Schizophrenia
Acronym: ASPIRE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 31-10-270
Record Dates: First submitted 2010-05-22; First posted 2010-05-25 (Estimated); Results first posted 2020-01-06 (Actual); Last update posted 2020-01-06 (Actual); Status verified 2019-12

CONDITIONS: Schizophrenia
Keywords: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Aripiprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Aripiprazole IM depot (Experimental): Active treatment of monthly doses of aripiprazole IM depot (300 mg or 400 mg)
  Interventions: Drug: Aripiprazole

INTERVENTIONS:
Drug: Aripiprazole — Aripiprazole IM depot - 300 mg or 400 mg

SUMMARY:
The primary objective of this study was to continue to provide aripiprazole intramuscular (IM) depot treatment (400 milligrams [mg] or 300 mg) to participants with schizophrenia completing the 52-week, open-label safety and tolerability Study 31-08-248. In addition, the secondary objective was to collect additional long-term safety data on aripiprazole IM depot treatment.

DETAILED DESCRIPTION:
This was an open-label study that enrolled participants with schizophrenia who had completed the 52-week, open-label safety and tolerability Study 31-08-248 and continued to provide aripiprazole IM depot treatment.

Participants received this treatment until aripiprazole IM Depot was commercially available in any dosage (including generic formulations) in the country where the study was being conducted or the commercial availability of aripiprazole IM Depot was terminated by the sponsor, or until the study completion date of 06 Dec 2018 was reached.

Eligible participants entered this study at the end of treatment visit (Week 52) of Study 31-08-248. Participants continued to receive aripiprazole IM depot every month (study months were every 4 weeks, which were defined as 28 [-2/+10] days) as a continuation of their previous monthly dose in Study 31-08-248.

ELIGIBILITY:
Inclusion Criteria:

* Participants with a current diagnosis of schizophrenia, as defined by Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition, Text Revision (DSM-IV-TR) criteria, who completed the open-label extension Study 248 (completed Study 248 study completion visit, Week 52).
* Participants who, in the investigator's judgment, may benefit from continued participation in an aripiprazole IM Depot study.
* The baseline visit for Study 270 (which is the Week 52 visit of Study 248) and the first injection for Study 270 must occur within 4 weeks (which was defined as 28 [-2/+10] days) of the last injection in Study 248.
* Participants who are able to provide written informed consent and/or consent obtained from a legally acceptable representative (as required by an Independent Review Board/Independent Ethics Committee (IRB/IEC), prior to the initiation of any protocol-required procedures.
* Participants able to understand the nature of the study and follow protocol requirements and who can read and understand the written word in order to complete patient-reported outcomes measures.
* Outpatient status.

Exclusion Criteria:

* Participants with a current DSM-IV-TR diagnosis other than schizophrenia, including schizoaffective disorder, major depressive disorder, bipolar disorder, delirium, dementia, amnestic, or other cognitive disorders.
* Participants with borderline, paranoid, histrionic, schizotypal, schizoid, or antisocial personality disorder.
* Participants who currently meet DSM-IV-TR criteria for substance dependence, including alcohol and benzodiazepines, but excluding caffeine and nicotine.
* Participants with a significant risk of violent behavior or a significant risk of committing suicide based on the investigator's judgment.
* Participants who are known to be allergic, intolerant, or unresponsive to prior treatment with aripiprazole or other quinolinones.
* Participants with a history of neuroleptic malignant syndrome or clinically significant tardive dyskinesia at screening.
* Electroconvulsive therapy within 180 days prior to entry.
* Any participant who requires or may need any other antipsychotic medications during the course of the study.
* Aripiprazole IM Depot (including generic formulation) is commercially available in the participant's country.
* Other protocol specific inclusion/exclusion criteria may apply.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 709 (Actual)
Dates: Start 2010-06-24 (Actual); Primary Completion 2018-12-06 (Actual); Study Completion 2018-12-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (129):
- United States (46):
  - Bellevue, California
  - Garden Grove, California
  - Glendale, California
  - Imperial, California
  - Los Angeles, California
  - National City, California
  - Orange, California
  - Pasadena, California
  - Pico Rivera, California
  - San Bernardino, California
  - San Diego, California
  - Sherman Oaks, California
  - Norwalk, Connecticut
  - Washington D.C., District of Columbia
  - Bradenton, Florida
  - Doral, Florida
  - Hialeah, Florida
  - Homestead, Florida
  - Orange City, Florida
  - Tampa, Florida
  - Chicago, Illinois
  - Oak Brook, Illinois
  - Indianapolis, Indiana
  - Shreveport, Louisiana
  - Flowood, Mississippi
  - St Louis, Missouri
  - North Platte, Nebraska
  - Buffalo, New York
  - New York, New York
  - Queens, New York
  - Rochester, New York
  - Charlotte, North Carolina
  - Akron, Ohio
  - Canton, Ohio
  - Toledo, Ohio
  - Oklahoma City, Oklahoma
  - Allentown, Pennsylvania
  - Jenkintown, Pennsylvania
  - Sellersville, Pennsylvania
  - Charleston, South Carolina
  - Memphis, Tennessee
  - Austin, Texas
  - DeSoto, Texas
  - Richmond, Virginia
  - Bothell, Washington
  - Milwaukee, Wisconsin
- Argentina (2):
  - Buenos Aires
  - Mendoza
- Australia (3):
  - Epping, Victoria
  - Frankston, Victoria
  - Fremantle, Western Australia
- Bulgaria (10):
  - Burgas
  - Lovech
  - Pazardzhik
  - Pleven
  - Plovdiv
  - Radnevo
  - Rousse
  - Sofia
  - Tserova Koria
  - Varna
- Chile (3):
  - Santiago
  - Temuco
  - Valdivia
- Zagreb, Croatia
- Estonia (3):
  - Tallinn
  - Tartu
  - Viljandi
- Helsinki, Finland
- Hungary (3):
  - Baja
  - Balassagyarmat
  - Gyõr
- India (7):
  - Ahmedabad, Gujarat
  - Mangalore, Karnataka
  - Bangalore
  - Chennai
  - Kanpur
  - Pune
  - Tirupati
- Malaysia (3):
  - Ipoh
  - Kajang
  - Kuala Lumpur
- Mexico (5):
  - Guadalajara, Jalisco
  - Monterrey, Nuevo León
  - Culiacán, Sinaloa
  - México
  - San Luis Potosí City
- Philippines (3):
  - Mandaluyong, NCR
  - Iloilo City, Western Visayas
  - Mariveles
- Poland (8):
  - Bełchatów
  - Bialystok
  - Bydgoszcz
  - Choroszcz
  - Krakow
  - Leszno
  - Sosnowiec
  - Wroclaw
- San Juan, Puerto Rico
- Romania (6):
  - Arad
  - Bucharest
  - Cluj-Napoca
  - Craiova
  - Oradea
  - Piteşti
- Russia (5):
  - Lipetsk
  - Moscow
  - Nizhny Novgorod
  - Saint Petersburg
  - Smolensk
- Serbia (2):
  - Belgrade
  - Kragujevac
- Slovakia (5):
  - Bardejov
  - Košice
  - Liptovský Mikuláš
  - Prešov
  - Rimavská Sobota
- South Africa (3):
  - Cape Town, Western Province
  - Bellville
  - Pretoria West
- South Korea (4):
  - Daejeon
  - Gwangju
  - Incheon
  - Seoul
- Spain (2):
  - Barcelona
  - L'Hospitalet de Llobregat
- Taiwan (2):
  - Tainan
  - Taipei
- Chiang Mai, Thailand

IPD SHARING:
Plan to Share IPD: Yes
Anonymized Individual participant data (IPD) that underlie the results of this study will be shared with researchers to achieve aims pre-specified in a methodologically sound research proposal. Small studies with less than 25 participants are excluded from data sharing.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data will be available after marketing approval in global markets, or beginning 1-3 years following article Publication. There is no end date to the availability of the data.
Access Criteria: Otsuka will share data on an Otsuka-owned remotely accessible data sharing platform with Python and R analytical software. Research requests should be directed to clinicaltransparency@Otsuka-us.com.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants with a current diagnosis of schizophrenia, as defined by Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition, Text Revision (DSM-IV-TR) criteria, who completed the open-label extension Study 31-08-248 (NCT00731549) (completed Study 248 Study Completion visit, Week 52).
Groups:
- Aripiprazole IM Depot: Monthly dose of 400 milligrams (mg) or 300 mg aripiprazole intramuscular (IM) depot to adult participants with schizophrenia who completed aripiprazole IM depot treatment in Study 31-08-248.
Period: Overall Study
Arm/Group | Aripiprazole IM Depot
Started | 709
Received at Least 1 Dose of Study Drug | 709
Completed | 431
Not Completed | 278
Not completed — Adverse Event | 39
Not completed — Death | 6
Not completed — Lack of Efficacy | 5
Not completed — Lost to Follow-up | 13
Not completed — Physician Decision | 27
Not completed — Protocol Deviation | 3
Not completed — Withdrawal Criteria Met | 19
Not completed — Trial Termination by Sponsor | 6
Not completed — Withdrawal by Subject | 160

BASELINE CHARACTERISTICS:
Population: All participants who completed week 52 of Study 31-08-248 and enrolled in Study 31-10-270.
Arm/Group | Aripiprazole IM Depot
Number analyzed (Participants) | 709
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 709
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: Years]
  Age (years) | 41.9 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 295
  Male | 414
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 464
  Black or African American | 78
  American Indian or Alaska Native | 1
  Asian | 107
  Native Hawaiian or Other Pacific Islander | 1
  Other | 58

OUTCOME MEASURES:

1. Primary Outcome: Number Of Participants Reporting Severe Treatment-Emergent Adverse Events (TEAE)
Description: A TEAE was defined as an AE that started after start of investigational medicinal product (IMP) treatment or if the event was continuous from baseline and was serious, IMP-related, or resulted in death, discontinuation, interruption, or reduction of IMP. A severe AE was one that caused inability to work or perform normal daily activity.
  A summary of serious and all other non-serious adverse events, regardless of causality, is located in the Reported Adverse Events module.
Time Frame: Baseline to Month 97 (+/- 3 days)
Population: The Safety Sample includes all participants who received at least 1 dose of open-label aripiprazole IM depot.
Measure: Number; unit: participants
Arm/Group | Aripiprazole IM Depot
Number analyzed (Participants) | 709
participants | 50

2. Secondary Outcome: Mean Change In Clinical Global Impression-Severity (CGI-S) of Illness Scale Score From Baseline To Last Visit
Description: The severity of illness for each participant was rated using the CGI-S scale. To assess CGI-S, the rater or investigator answered the following question: "Considering your total clinical experience with this particular population, how mentally ill is the patient at this time?" Response choices included: 0 = not assessed; 1 = normal, not ill at all; 2 = borderline mentally ill; 3 = mildly ill; 4 = moderately ill; 5 = markedly ill; 6 = severely ill; and 7 = among the most extremely ill patients. The Last Visit was defined as the last available post-baseline evaluation. A decrease in the CGI-S score indicated disease stability or improvement.
Time Frame: Baseline, Month 91
Population: The Efficacy Sample comprises those participants who entered the trial and had at least 1 post-baseline efficacy evaluation.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Aripiprazole IM Depot
Number analyzed (Participants) | 703
units on a scale | -0.14 (0.69)

ADVERSE EVENTS:
Time Frame: Baseline to Month 97 (+/- 3 days)
Description: The Safety Sample comprised all participants who received at least 1 dose of open-label aripiprazole IM depot.
Arm/Group | Aripiprazole IM Depot
All-Cause Mortality (participants affected / at risk) | 6/709
Serious Adverse Events (participants affected / at risk) | 62/709
Other Adverse Events (participants affected / at risk) | 515/709
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aripiprazole IM Depot (N=709)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
Supraventricular Tachycardia (Cardiac disorders) | 1 (1)
Acute Myocardial Infarction (Cardiac disorders) | 1 (1)
Arteriospasm Coronary (Cardiac disorders) | 1 (1)
Myocardial Ischaemia (Cardiac disorders) | 1 (1)
Cardio-Respiratory Arrest (Cardiac disorders) | 1 (1)
Vitello-Intestinal Duct Remnant (Congenital, familial and genetic disorders) | 1 (1)
Death (General disorders) | 1 (1)
Hepatic Failure (Hepatobiliary disorders) | 1 (1)
Autoimmune Hepatitis (Hepatobiliary disorders) | 1 (1)
Hepatic Cirrhosis (Hepatobiliary disorders) | 1 (1)
Pneumonia Bacterial (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 3 (3)
Oesophageal Candidiasis (Infections and infestations) | 1 (1)
Influenza (Infections and infestations) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 1 (1)
Pulmonary Tuberculosis (Infections and infestations) | 1 (1)
Infection (Infections and infestations) | 1 (1)
Erysipelas (Infections and infestations) | 1 (1)
Abscess Jaw (Infections and infestations) | 1 (1)
Abdominal Abscess (Infections and infestations) | 1 (1)
Abdominal Infection (Infections and infestations) | 1 (1)
Dengue Fever (Infections and infestations) | 1 (1)
Bacteraemia (Infections and infestations) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1)
Accidental Overdose (Injury, poisoning and procedural complications) | 1 (1)
Gun Shot Wound (Injury, poisoning and procedural complications) | 1 (1)
Foot Fracture (Injury, poisoning and procedural complications) | 1 (1)
Road Traffic Accident (Injury, poisoning and procedural complications) | 1 (1)
Hepatic Enzyme Increased (Investigations) | 1 (1)
Type 2 Diabetes Mellitus (Metabolism and nutrition disorders) | 1 (1)
Diabetes Mellitus (Metabolism and nutrition disorders) | 1 (1)
Haemosiderosis (Metabolism and nutrition disorders) | 1 (1)
Still's Disease (Musculoskeletal and connective tissue disorders) | 1 (1)
Pancreatic Carcinoma Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Cerebellar Tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Lung Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Metastases to Liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Pleomorphic Adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Presyncope (Nervous system disorders) | 1 (1)
Cerebrovascular Accident (Nervous system disorders) | 1 (1)
Thrombotic Cerebral Infarction (Nervous system disorders) | 1 (1)
Seizure (Nervous system disorders) | 2 (2)
Loss of Consciousness (Nervous system disorders) | 1 (1)
Psychotic Disorder (Psychiatric disorders) | 9 (9)
Suicide Attempt (Psychiatric disorders) | 2 (2)
Suicidal Behaviour (Psychiatric disorders) | 1 (1)
Schizophrenia (Psychiatric disorders) | 14 (14)
Insomnia (Psychiatric disorders) | 1 (1)
Aggression (Psychiatric disorders) | 1 (1)
Delusion (Psychiatric disorders) | 1 (1)
Acute Stress Disorder (Psychiatric disorders) | 1 (1)
Suicidal Ideation (Psychiatric disorders) | 1 (1)
Impulse-Control Disorder (Psychiatric disorders) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1)
Cystocele (Reproductive system and breast disorders) | 1 (1)
Metrorrhagia (Reproductive system and breast disorders) | 1 (1)
Ovarian Cyst (Reproductive system and breast disorders) | 1 (1)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary Hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Skin Ulcer (Skin and subcutaneous tissue disorders) | 1 (1)
Dermatitis Allergic (Skin and subcutaneous tissue disorders) | 1 (1)
Poor Personal Hygiene (Social circumstances) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aripiprazole IM Depot (N=709)
Diarrhoea (Gastrointestinal disorders) | 37 (37)
Influenza (Infections and infestations) | 48 (48)
Nasopharyngitis (Infections and infestations) | 87 (87)
Upper Respiratory Tract Infection (Infections and infestations) | 54 (54)
Weight Increased (Investigations) | 81 (81)
Back Pain (Musculoskeletal and connective tissue disorders) | 42 (42)
Headache (Nervous system disorders) | 77 (77)
Anxiety (Psychiatric disorders) | 44 (44)
Insomnia (Psychiatric disorders) | 70 (70)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right to review results publications prior to public release and can delay such publications for a period greater than 60 days but no more than 120 days from the date that the publication is submitted to the Sponsor for review. Sponsor can require changes to the publication to protect Sponsor's intellectual property rights and/or confidential information and reserves the right to limit publication timing and scope of data published based on the number of study locations.

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-12-12): https://cdn.clinicaltrials.gov/large-docs/82/NCT01129882/SAP_000.pdf
  • Study Protocol (2015-07-08): https://cdn.clinicaltrials.gov/large-docs/82/NCT01129882/Prot_001.pdf